CLINICAL TRIAL: NCT00002332
Title: Double-Blind Study of the Effect of Timunox (Thymopentin) on Lymphoproliferative Responses and Virus Load in HIV-Infected Subjects Receiving Nucleoside Analog Antiretroviral Therapy
Brief Title: A Study of Timunox (Thymopentin) in HIV-Infected Patients Receiving Other Anti-HIV Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immunobiology Research Institute (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 015I; 07.32.039-94
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-12

CONDITIONS: HIV Infections
Keywords: Thymopentin; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Thymopentin

INTERVENTIONS:
Drug: Thymopentin

SUMMARY:
To evaluate the mechanism whereby thymopentin appears to retard the progressive immune suppression attributable to HIV infection.

DETAILED DESCRIPTION:
Patients are randomized to receive subcutaneous thymopentin or placebo thrice weekly for 4 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Asymptomatic or minimally symptomatic HIV infection (no evidence of AIDS).
* CD4 count <= 400 cells/mm3 within 6 weeks prior to study entry (CD4 count changed to 100 - 400 cells/mm3 per amendment).
* Tolerated the current nucleoside analog antiretroviral treatment for at least 4 weeks prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known hypersensitivity to thymopentin or any component of the formulation.
* Significant chronic underlying medical illness that would impede study participation.
* Grade 2 or higher peripheral neuropathy related to nucleoside analog antiretroviral treatment.

Concurrent Medication:

Excluded:

* Any antiretroviral agents other than zidovudine, didanosine, or dideoxycytidine.
* HIV vaccines or any investigational or non-FDA approved medication or immunomodulatory or experimental therapy within 30 days prior to study entry.

Patients with the following prior condition are excluded:

Abnormal chest x-ray consistent with active opportunistic infection within 6 weeks prior to study entry.

Prior Medication:

Excluded:

* Any prior antiretroviral agents other than zidovudine, didanosine, or dideoxycytidine within 30 days prior to study entry.

Required:

* Current nucleoside analog antiretroviral treatment.

Required:

* Nucleoside analog antiretroviral treatment for at least 4 weeks prior to study entry.

Significant active alcohol or drug abuse sufficient to prevent study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Dr Marcus Conant, San Francisco, California
  - Dr Jeffrey Galpin, Tarzana, California
  - Novum Inc, Pittsburgh, Pennsylvania